CLINICAL TRIAL: NCT00498368
Title: A Multicenter, Randomized, Prospective, Open-Label Trial of Rituximab in the Treatment of Progressive IgA Nephropathy
Brief Title: Rituximab in Progressive Immunoglobulin A (IgA) Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Ohio State University (Other); Stanford University (Other); University of North Carolina, Chapel Hill (Other); Columbia University (Other); Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Fernando Fervenza, M.D., Ph.D, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-001944
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: IgA Nephropathy
Keywords: Estimated glomerular filtration rate (GFR); Proteinuria; Renal Fibrosis
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab Plus ACE/ARB (Experimental): Intravenous Rituximab therapy, ACE/ARB combination therapy, and Omega-3 Fatty Acid Fish Oil Supplement
  Interventions: Drug: Intravenous Rituximab; Drug: ACE/ARB; Dietary Supplement: Omega-3 Fatty Acid Fish Oil Supplement
- ACE/ARB (Active Comparator): ACE/ARB therapy and Omega-3 Fatty Acid Fish Oil Supplement
  Interventions: Drug: ACE/ARB; Dietary Supplement: Omega-3 Fatty Acid Fish Oil Supplement

INTERVENTIONS:
Drug: Intravenous Rituximab — Rituximab Therapy [27 Patients]
  * Rituximab 1 gm IV on Treatment Day 1
  * Rituximab 1 gm IV on Treatment Day 15
  * Rituximab 1 gm IV on Treatment Day 168
  * Rituximab 1 gm IV on Treatment Day 182
  Other Names: Rituxan
  Arms: Rituximab Plus ACE/ARB
Drug: ACE/ARB — ACE inhibitors and /or ARBs will be used to achieve a blood pressure goal of <130/80 millimeters of mercury (mmHg). Patients not attaining the target blood pressure with an ACE inhibitor or ARB alone should be treated with the combination of ACE inhibitor (ACEi) + ARB
  Other Names: Angiotensin II blockade
Dietary Supplement: Omega-3 Fatty Acid Fish Oil Supplement — Omega-3 Fatty Acid Fish Oil Supplement 3.6 gm eicosapentaenoic acid (EPA)/day

SUMMARY:
This study was about IgA nephropathy, a form of kidney disease characterized by the presence of blood and protein in the urine. This study was done to determine if the medication rituximab could reduce protein in the patient's urine.

Hypothesis: In patients with progressive IgA nephropathy an intravenous infusion of 1000 mg of rituximab on Day 1 and Day 15 and Days 168 and 182 is superior to conventional therapy in reducing 24 hour proteinuria, and slowing progression of chronic kidney disease.

DETAILED DESCRIPTION:
Recent clinical success in the use of Rituximab in the treatment of Lupus nephritis and other forms immune complex glomerulonephritis has led to its investigation in the treatment of IgA nephropathy. Because IgA class antibodies have comparatively short half-lives and that deposition of polymeric forms of IgA contributes to glomerular injury, the researchers speculated that the reduction of circulating IgA could reduce proteinuria and injury in patients with IgA nephropathy.

Treatment and Follow-up:

Subjects were randomly assigned to receive rituximab or to continue standard care. Both arms received a Omega-3 Fatty Acid Fish Oil Supplement and angiotensin converting enzyme (ACE) inhibitors and/or Angiotensin II receptor blockers (ARBs). ACE inhibitors and/or ARBs were used to achieve a blood pressure goal of <130/80 mmHg.

The study was an open-label trial; those assigned to rituximab received a 1 g infusion of rituximab followed by an identical dose 2 weeks later. Premedication with corticosteroids (10 mg dexamethasone intravenously) was also given 30 min prior to the first infusion of each series of rituximab. They received an identical 2 g course of rituximab 6 months later. Subjects were assessed at least every 3 months or as needed for clinical events. This assessment included physical examination, a questionnaire for adverse events, and measurement of routine hematology, serum chemistry, timed urine protein excretion, and for those assigned to rituximab, B-cell subsets. Follow-up was considered complete at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Any patient between the age of 18 and 70 years of age and able to give informed consent
* GFR by Cockcroft-Gault or MDRD equations <90 mls/min and >30 mls/min
* Greater than or equal to 1000 mg of proteinuria/24 hours while on stable ACEi, ARB or renin inhibitor therapy for 2 months. Patients receiving combination ACE or ARB or ACEi and a renin inhibitor for 2 months will only require 500mg/24 hours
* Blood pressure <130/80 mmHg. The presence of hypertension is not required for study entry, but any patient requiring long term hypertensive medications must have blood pressure controlled <130-80 mmHg, to be considered eligible for the study
* Female patients with IgA will be considered eligible for study entry if they have a negative urine or serum pregnancy test at the time of screening are agreeable to 2 years of contraception
* Biopsy proven IgA nephropathy and clinical features consistent with Henoch Schonlein Purpura will be considered eligible for the study
* Able to swallow the oral medications

Exclusion Criteria

* Clinical and histologic evidence of IgA predominant Lupus nephritis
* Clinical and histologic evidence of idiopathic IgA forms of membranoproliferative glomerulonephritis
* Clinical evidence of cirrhosis, chronic active liver disease or known infection with hepatitis B, C or HIV
* Estimated GFR <30 ml/min/1.73m² at the time of screening
* Greater than 50% glomerular senescence or cortical scarring on renal biopsy
* Active systemic infection or history of serious infection within one month of entry
* History of Crohn's disease or Celiac Sprue
* Positive pregnancy test or breast feeding at time of study entry or unwilling to comply with contraceptive measures
* Current or recent (within 30 days) exposure to any investigational drug
* Serum Cr >3.5 mg/dl or Modification of Diet in Renal Disease (MDRD) calculated GFR <30 mls/min
* Patients receiving >6 months therapy with oral prednisone or glucocorticoid equivalent
* Live vaccine within 28 days of study enrollment.

General Safety & Laboratory Exclusion Criteria

* Patients with anaphylaxis and/or known allergic reactions to Rituximab
* Hemoglobin: <8.5 gm/dL
* Platelets: <100,000/mm
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 x Upper Limit of Normal unless related to primary disease.
* Previous Treatment with Rituximab(MabThera®/Rituxan®)
* Previous treatment with Natalizumab(Tysabri®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent significant infection or recurrent bacterial infections
* Known active bacterial, viral fungal mycobacterial or atypical mycobacterial infections, but excluding fungal infections of nail beds
* Any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Ongoing use of high dose steroids(>10 mg/day)or unstable steroid dose in the past 4 weeks
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum or urine pregnancy test will be performed for all women of childbearing potential no later than 7 days prior to treatment) or lactation
* Concomitant or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complication
* Inability to comply with study and follow-up procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C. Fervenza, M.D., Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Stanford University, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - The University of Ohio, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lafayette RA, Canetta PA, Rovin BH, Appel GB, Novak J, Nath KA, Sethi S, Tumlin JA, Mehta K, Hogan M, Erickson S, Julian BA, Leung N, Enders FT, Brown R, Knoppova B, Hall S, Fervenza FC. A Randomized, Controlled Trial of Rituximab in IgA Nephropathy with Proteinuria and Renal Dysfunction. J Am Soc Nephrol. 2017 Apr;28(4):1306-1313. doi: 10.1681/ASN.2016060640. Epub 2016 Nov 7. PMID 27821627
- [Derived] Yeo SC, Liew A, Barratt J. Emerging therapies in immunoglobulin A nephropathy. Nephrology (Carlton). 2015 Nov;20(11):788-800. doi: 10.1111/nep.12527. PMID 26032537

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Plus ACE/ARB: Intravenous Rituximab therapy, ACE/ARB combination therapy, and Omega-3 Fatty Acid Fish Oil Supplement
  Intravenous Rituximab: Rituximab Therapy [27 Patients]
  * Rituximab 1 gm IV on Treatment Day 1
  * Rituximab 1 gm IV on Treatment Day 15
  * Rituximab 1 gm IV on Treatment Day 168
  * Rituximab 1 gm IV on Treatment Day 182
  * An angiotensin converting enzyme (ACE) inhibitors and /or angiotensin II receptor blockers (ARBs) will be used to achieve a B/P goal of <130/80 millimeters of mercury
  Omega-3 Fatty Acid Fish Oil Supplement: Omega-3 Fatty Acid Fish Oil Supplement 3.6 gm eicosapentaenoic acid (EPA)/day
- ACE/ARB: ACE/ARB therapy and Omega-3 Fatty Acid Fish Oil Supplement
  ACE/ARB: ACE inhibitors and /or ARBs will be used to achieve a B/P goal of <130/80 millimeters of mercury (mmHg)
  Omega-3 Fatty Acid Fish Oil Supplement: Omega-3 Fatty Acid Fish Oil Supplement 3.6 gm eicosapentaenoic acid (EPA)/day
Period: Overall Study
Arm/Group | Rituximab Plus ACE/ARB | ACE/ARB
Started | 17 | 17
Completed | 14 | 15
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rituximab Plus ACE/ARB: Intravenous Rituximab therapy, ACE/ARB combination therapy, and Omega-3 Fatty Acid Fish Oil Supplement
  Intravenous Rituximab: Rituximab Therapy [27 Patients]
  * Rituximab 1 gm IV on Treatment Day 1
  * Rituximab 1 gm IV on Treatment Day 15
  * Rituximab 1 gm IV on Treatment Day 168
  * Rituximab 1 gm IV on Treatment Day 182
  * An ACE inhibitors and /or ARBs will be used to achieve a blood pressure goal of <130/80 millimeters of mercury (mmHg)
  Omega-3 Fatty Acid Fish Oil Supplement: Omega-3 Fatty Acid Fish Oil Supplement 3.6 gm eicosapentaenoic acid (EPA)/day
- ACE/ARB: ACE/ARB therapy and Omega-3 Fatty Acid Fish Oil Supplement
  ACE/ARB: ACE inhibitors and /or ARBs will be used to achieve a blood pressure goal of <130/80 millimeters of mercury (mmHg)
  Omega-3 Fatty Acid Fish Oil Supplement: Omega-3 Fatty Acid Fish Oil Supplement 3.6 gm eicosapentaenoic acid (EPA)/day
- Total: Total of all reporting groups
Arm/Group | Rituximab Plus ACE/ARB | ACE/ARB | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Median (Full Range); unit: years] | 43 [29 to 63] | 33 [21 to 59] | 40 [21 to 63]
Gender [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 10 | 15 | 25
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Proteinuria at 12 Months
Time Frame: 1 year
Population: The number of participants differs from the participant flow because not all participants had the laboratory test done.
Measure: Number; unit: participants
Arm/Group | Rituximab Plus ACE/ARB | ACE/ARB
Number analyzed (Participants) | 10 | 10
participants
  Number of participants with > 50% reduction | 3 | 3
  Number of participants with >50% increase | 1 | 2
  Number of participants with <500 mg of protein | 2 | 2

2. Secondary Outcome: Biochemical Marker IgA at 12 Months
Time Frame: 12 months
Population: The number of participants differs from the participant flow because not all participants had the laboratory test done.
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Rituximab Plus ACE/ARB | ACE/ARB
Number analyzed (Participants) | 10 | 10
mg/ml | 4.4 (1.4) | 4.6 (1.9)

3. Secondary Outcome: Biochemical Marker Gd-Immunoglobulin A Subclass 1 (IgA1) at 12 Months
Time Frame: 12 months
Population: The number of participants differs from the participant flow because not all participants had the laboratory test done.
Measure: Mean (Standard Deviation); unit: U/100ng IgA
Arm/Group | Rituximab Plus ACE/ARB | ACE/ARB
Number analyzed (Participants) | 10 | 10
U/100ng IgA | 60.5 (13.0) | 58.9 (5.6)

4. Secondary Outcome: Biochemical Marker Immunoglobulin G (IgG) AutoAb at 12 Months
Time Frame: 12 months
Population: The number of participants differs from the participant flow because not all participants had the laboratory test done.
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Rituximab Plus ACE/ARB | ACE/ARB
Number analyzed (Participants) | 10 | 10
U/ml | 1751.3 (2469.4) | 1075 (908.7)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Rituximab Plus ACE/ARB | ACE/ARB
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No